CLINICAL TRIAL: NCT00580255
Title: Does Elevated Brain Natriuretic Peptide (BNP) Reflect Changes in Thoracic Impedance Levels and Affect Occurrence of Atrial and Ventricular Arrhythmias?
Brief Title: Comparison Study of BNP and Thoracic Impedance Measurements on Arrhythmias
Status: Withdrawn | Type: Observational
Why Stopped: resources not available
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200614766
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2013-01

CONDITIONS: Heart Failure; Arrhythmias
Keywords: CHF; CRT; Atrial Arrhythmias; Ventricular Arrhythmias; BioZ; Optivol
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Teaspoon of blood drawn for testing of BNP levels.
Oversight: Data Monitoring Committee: No

SUMMARY:
It is hypothesized that elevated BNP level correlate with an elevated thoracic impedance/fluid index as measured separately by CRT-D devices and external impedance cardiography. Ultimately, it is also hypothesized that both BNP and thoracic impedance/fluid index measurements are predictive of atrial and ventricular arrhythmias.

DETAILED DESCRIPTION:
The primary aim of this study:

1. To assess the correlation between elevated brain natriuretic peptide levels and elevated thoracic impedance/body fluid index as measured by selective biventricular resynchronization devices and an external impedance cardiography device.
2. Correlate impedance measurements and brain natriuretic levels with occurrence of atrial and ventricular arrhythmias as assessed by interrogation of biventricular devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 85 years of age.
* All patients with biventricular implantable cardio-defibrillators(manufacturer: Medtronic/ model: InSync 7299/7297 or newer).
* LVEF <35%
* NYHA III/IV
* QRS >120 msec
* Pt willing and able to sign informed consent.
* Conventional heart failure therapy
* Clinically stable for six months.

Exclusion Criteria:

* age less than 18 years of age
* age greater than 85 years of age
* Creatinine > 2.5 mg/dl.
* End stage liver disease complicated by ascites as determined by electronic medical record review.
* women who are pregnant, lactating, or plan to become pregnant during the course of the study.
* Patients who are heart transplant candidates with expected transplantation within the next six months.
* Life expectancy due to non-cardiac cause less than one year.
* Anticipated problem with compliance.
* Critical valvular stenoses/insufficiencies.
* Morbidly obese patients(>300 lbs.)
* In patients whom impedance cardiography was not able to be performed because of inability to place sensors.
* Planned or known need for revascularization procedures within three months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential candidates with criteria for implantable cardiac resynchronization therapy who have or will undergo implantation of a Medtronic CRT-D device with thoracic impedance measurement capabilities, will be eligible to enter the study if they meet all of the inclusion criteria and none of the exclusion criteria. Patients will be enrolled in the study either at the time of device implantation or if they have already undergone device implantation will be enrolled at next routine outpatient clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srivatsa, MD, Principal Investigator — U C Davis Medical Center
Locations (1):
- U C Davis Medical Center, Sacramento, California, United States